CLINICAL TRIAL: NCT01182961
Title: Gait Training Intervention to Evaluate the Efficacy of Using Virtual Reality to Decrease Fall Risk in the Elderly Population
Brief Title: The Use of Virtual Reality for the Gait Training of Elderly Fallers
Acronym: VR-Fallers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Nir Giladi, MD, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-10-NG-0113-CTIL
Record Dates: First submitted 2010-07-20; First posted 2010-08-17 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Elderly
Keywords: Gait; Falls; Virtual reality
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treadmill +virtual reality training (Experimental)
  Interventions: Other: gait training
- Treadmill alone (Active Comparator)
  Interventions: Other: gait training 2
- standard of care exercise group (Active Comparator)
  Interventions: Other: exercise group

INTERVENTIONS:
Other: gait training — subjects will walk on a treadmill while virtual obstacles will be displayed using a head mounted device
  Other Names: virtual reality
  Arms: Treadmill +virtual reality training
Other: gait training 2 — subjects will walk on a treadmill under a progressive intensive gait protocol
  Other Names: treadmill
  Arms: Treadmill alone
Other: exercise group — standard of care exercise group to improve strength and balance
  Arms: standard of care exercise group

SUMMARY:
The study aims to investigate the efficacy of gait training using virtual reality to decrease the risk of falls in elderly idiopathic fallers. The investigator hypothesize that training with virtual reality would increase the ability to perform in the "real world" environment and decrease the risk of falls in elderly adults.

DETAILED DESCRIPTION:
The study is a prospective single-blinded randomized control study with repeated measures at pre intervention, post intervention and follow up at 3 and 6 months post intervention. For six months after termination of the intervention, all subjects will fill out a log book in which they will write the occurrence and date of falls. total time of participation in the study will be 8 months.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 65-85
* independent in activities of daily living
* able to walk without assistance for at least 10 minutes
* cognitively intact (Mini Mental State Exam ≥24)
* reported 2 or more falls within 6 months prior to the beginning of the study

Exclusion Criteria:

* any neurological, orthopedic or any other impairment likely to impact gait.
* severe visual impairments
* major depression as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-09 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Gait dynamics | one week after training
  using an accelerometer, the coefficient of variation will be calculated

SECONDARY OUTCOMES:
cognitive function | one week after training
  using a cmputerized cognitive battary and neuropsychological testing

CONTACTS AND LOCATIONS:
Overall Officials: Nir Giladi, MD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel